CLINICAL TRIAL: NCT04967222
Title: Cognitive Reappraisal Training Targeting Emotion Circuits As a Therapeutic Intervention in Borderline Patients
Brief Title: Cognitive Reappraisal Training for Borderline Personality
Acronym: BPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: William Marsh Rice University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Harold W Koenigsberg, MD, Professor of Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-0432-01001; R61MH125130 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Borderline Personality Disorder
Keywords: BPD; Treatment; fMRI; cognitive reappraisal; Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Reappraisal-by-Distancing (CRD) (Experimental): Subjects will be coached to use cognitive reappraisal-by-distancing to downregulate their negative reactions to aversive emotional pictures usng practice pictures.
  Interventions: Behavioral: Cognitive Reappraisal by Distancing
- Control Downregulate Condition (CD) (Active Comparator): Subjects will be coached to practice their customary emotion regulatory techniques in a treatment occurring twice a week for 6 weeks.
  Interventions: Behavioral: Control Downregulate Condition

INTERVENTIONS:
Behavioral: Cognitive Reappraisal by Distancing — Reappraisal-by-distancing treatment. Participants meet 2 times a week for 6 weeks to learn reappraisal by distancing through repeated practice with negative emotional pictures. The therapist will help model and shape the technique. .
  Other Names: CRD
  Arms: Cognitive Reappraisal-by-Distancing (CRD)
Behavioral: Control Downregulate Condition — Participants either meet 2x a week for 6- weeks to gain added practice, under the guidance of a therapist, using their customary emotion regulatory strategies to downregulate their negative reactions to aversive pictures.
  Other Names: CD
  Arms: Control Downregulate Condition (CD)

SUMMARY:
Previous work by the study group convinced the study team to pursue development of focused cognitive reappraisal training as a novel approach to treatment of BPD, either as stand-alone treatment or in concert with evidence-based treatments of BPD. The present proposal aims to refine and test a proposed clinical intervention for BPD patients, training in reappraisal-by-distancing, in terms of its ability to influence hypothesized neural and behavioral targets and, once that is established, to demonstrate its ability improve clinically relevant outcome measures.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a prevalent, enduring and disabling psychiatric condition found in approximately 2% to 5.9% of the population and 20% of hospitalized psychiatric patients. Suicide rates of approximately 10% have been reported. One of the most prominent clinical features of BPD is extreme mood shifts occurring in response to external social/emotional events. The emotional instability in BPD contributes to many of the most disabling, even life-threatening, symptoms of the disorder, including suicidality, outbursts of intense anger, and seriously impaired role functioning. The severity of the BPD symptom profile, its prevalence, chronicity and high burden upon health care services make the development of effective and accessible treatment for BPD a high priority. Yet there is no current medication treatment indicated for BPD and the psychotherapies recognized for the disorder have been shown to have small effect sizes and are of limited availability.

The present study builds upon work by the study group that has shown that deficiencies in the ability to regulate emotion by engaging typically adaptive cognitive strategies (cognitive reappraisal, CR) and to effectively activate associated neural systems can be corrected by focused training in CR. The R61 phase of this study examines a manualized intensive training program in CR, tests that it effects target neural systems implicated in emotional processing and enhances behavioral reappraisal success. It examines 2-, 4- and 6- weeks of twice a week treatment to identify the optimal dose. Measures include fMRI imaging and clinical ratings at baseline and each of these subsequent time points. Upon demonstrating that CR training is superior to a control condition in enhancing performance in the neural target at one or more of these dose durations, the study team will proceed to the R33 phase. In the R33 phase the study team will treat a larger sample of BPD patients at the optimal dose defined in the R61 phase to 1) demonstrate reproducibility of the R61 findings, 2) to demonstrate that CR training is superior to control in improving BPD clinical outcomes at the end of treatment and at 1- and 4- month follow-up, and 3) that change in activity at the neural targets is associated with clinical improvement.

The results of this study can support the introduction of CR training as a new psychosocial approach for the treatment of BPD, either as stand-alone treatment or as an augmenting strategy. It may, moreover, have application to a range of psychiatric disorders characterized by severe emotional instability.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy men and women with Borderline Personality Disorder who are mentally competent and give informed voluntary written consent.
* Subjects who are being treated with psychotherapy or psychopharmacotherapy will be included so long as there has been no change in that treatment over the preceding 2 months.

Exclusion Criteria:

* Age > 55
* Criteria for Schizotypal Personality Disorder or Avoidant Personality Disorder. SPD is excluded to avoid possible confound from the restricted affect that characterizes SPD and co-morbid AvPD subjects will be excluded because the researchers have shown that their patterns of neural activity in emotion processing are distinct from BPD subjects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold Koenigsberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. For individual participant data meta-analysis.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 participants consented. After preliminary screening visits, 26 participants were randomized.
Groups:
- All Participants Consented: All participants consented and had screening visit
- Cognitive Reappraisal-by-Distancing (CRD): Subjects will be coached to use cognitive reappraisal-by-distancing to downregulate their negative reactions to aversive emotional pictures using practice pictures.
  Cognitive Reappraisal by Distancing: Reappraisal-by-distancing treatment. Participants meet 2 times a week for 6 weeks to learn reappraisal by distancing through repeated practice with negative emotional pictures. The therapist will help model and shape the technique.
Period: Screening Visits
Arm/Group | All Participants Consented | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Started | 60 | 0 | 0
Completed | 26 | 0 | 0
Not Completed | 34 | 0 | 0
Period: Randomized
Arm/Group | All Participants Consented | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Started | 0 | 13 | 13
Completed | 0 | 10 | 9
Not Completed | 0 | 3 | 4
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — abnormal finding in MRI | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.08 (8.14) | 30.46 (9.22) | 30.77 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 6 | 8 | 14
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in PINES Network Activity
Description: BOLD signal change in Picture Induced Negative Emotion Signature (PINES) network activity that includes the amygdala, insula, and other regions by measuring neural activation using fMRI.
Time Frame: Baseline and up to 6 weeks of treatment
Population: Data available for participants who had procedure
Measure: Mean (Standard Deviation); unit: BOLD Signal
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Number analyzed (Participants) | 13 | 13
BOLD Signal
  baseline: number analyzed (Participants) | 13 | 12
  baseline | 0.15 (0.04) | 0.14 (0.03)
  after up to 6 weeks of treatment: number analyzed (Participants) | 7 | 8
  after up to 6 weeks of treatment | 0.12 (0.04) | 012 (0.06)

2. Primary Outcome: Change in Zanarini Rating Scale for Borderline Personality (ZAN-BPD)
Description: Zanarini Rating Scale for Borderline Personality, self-report. Full scale from 0-36. Higher score indicates poorer health outcomes.
Time Frame: Baseline and up to 6 weeks of treatment
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline: number analyzed (Participants) | 9 | 7
  Baseline | 15.22 (7.70) | 12.86 (5.70)
  after up to 6 weeks of treatment: number analyzed (Participants) | 8 | 8
  after up to 6 weeks of treatment | 10 (9.52) | 9.38 (6.19)

3. Secondary Outcome: Change in ZAN-BPD Sector Scores
Description: There are three affective symptoms in the ZAN-BPD (with a sector score ranging from 0-12): inappropriate anger/frequent angry acts, mood instability, and chronic feelings of emptiness. There are two cognitive symptoms (with a sector score ranging from 0-8): stress-related paranoia/dissociation and severe identity disturbance. (Identity disturbance was placed in the cognitive realm because it is based on a series of false beliefs or overvalued ideas, such as that one is a bad person.) There are also two impulsive symptoms (with a sector score ranging from 0-8): self-mutilative/suicidal efforts and at least two other forms of impulsivity. Finally, there are two symptoms in the interpersonal realm of BPD (with a sector score ranging from 0-8): frantic efforts of avoid abandonment and intense, unstable relationships. The four sector scores sum to provide a total score of borderline psychopathology, which ranges from 0-36. Higher score indicates poorer health outcomes
Time Frame: Baseline and at 2-,4-, and 6-weeks
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline - Affective Sector: number analyzed (Participants) | 9 | 7
  Baseline - Affective Sector | 5.33 (2.29) | 5 (2.83)
  Baseline - Cognitive Sector: number analyzed (Participants) | 9 | 7
  Baseline - Cognitive Sector | 4 (2.45) | 2.71 (1.80)
  Baseline - Impulsive Sector: number analyzed (Participants) | 9 | 7
  Baseline - Impulsive Sector | 1.89 (1.83) | 2.57 (1.40)
  Baseline - Interpersonal Sector: number analyzed (Participants) | 9 | 7
  Baseline - Interpersonal Sector | 4 (2.24) | 2.57 (1.13)
  2 weeks - Affective Sector: number analyzed (Participants) | 10 | 10
  2 weeks - Affective Sector | 4.3 (3.13) | 4.5 (2.42)
  2 weeks - Cognitive Sector: number analyzed (Participants) | 10 | 10
  2 weeks - Cognitive Sector | 2.8 (2.49) | 2.1 (1.85)
  2 weeks - Impulsive Sector: number analyzed (Participants) | 10 | 10
  2 weeks - Impulsive Sector | 1.9 (1.91) | 1.3 (0.82)
  2 weeks- Interpersonal Sector: number analyzed (Participants) | 10 | 10
  2 weeks- Interpersonal Sector | 2.5 (2.37) | 2 (1.63)
  4 weeks - Affective Sector: number analyzed (Participants) | 7 | 4
  4 weeks - Affective Sector | 4 (2.89) | 2.75 (3.40)
  4 weeks - Cognitive Sector: number analyzed (Participants) | 7 | 4
  4 weeks - Cognitive Sector | 2.57 (2.76) | 1.75 (1.71)
  4 weeks - Impulsive Sector: number analyzed (Participants) | 7 | 4
  4 weeks - Impulsive Sector | 1.43 (2.15) | 0.75 (0.96)
  4 weeks - Interpersonal Sector: number analyzed (Participants) | 7 | 4
  4 weeks - Interpersonal Sector | 2.14 (2.34) | 2.25 (1.71)
  6 weeks - Affective Sector: number analyzed (Participants) | 8 | 8
  6 weeks - Affective Sector | 3.5 (3.42) | 4 (2.20)
  6 weeks - Cognitive Sector: number analyzed (Participants) | 8 | 8
  6 weeks - Cognitive Sector | 3.125 (2.8) | 2.13 (2.03)
  6 weeks - Impulsive Sector: number analyzed (Participants) | 8 | 8
  6 weeks - Impulsive Sector | 1.38 (2.00) | 1 (1.07)
  6 weeks - Interpersonal Sector: number analyzed (Participants) | 8 | 8
  6 weeks - Interpersonal Sector | 2.38 (2.50) | 2.5 (2.40)

4. Secondary Outcome: Change in Affective Lability Scale Total (ALS)
Description: The Affective Lability Scale (ALS) consists of 54 items which are rated on a four-point Likert scale ranging from 0 ("very uncharacteristic of me") to 3 ("very characteristic of me"). Five of the items refer to shifts in anxiety/depression, eight refer to shifts in depression/elation, and the final five items concern shifts between anger and normal mood. The scale yields a total score of ALS, as well as subscores for the three affective domains. Total score range from 0 to 162, with higher score indicating more affective lability.
Time Frame: Baseline and at 2-,4-, and 6-weeks
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline: number analyzed (Participants) | 13 | 12
  Baseline | 95 (25.52) | 104 (17.29)
  2 weeks: number analyzed (Participants) | 11 | 11
  2 weeks | 82.91 (26.11) | 93.27 (16.75)
  4 weeks: number analyzed (Participants) | 10 | 10
  4 weeks | 74.3 (32.67) | 85.8 (23.01)
  6 weeks: number analyzed (Participants) | 10 | 9
  6 weeks | 80.7 (38.21) | 87.11 (16.17)

5. Secondary Outcome: Change in Perceived Stress Scale (PSS)
Description: Perceive Stress Scale (PSS) - A 10-item questionnaire, each item scored 0 (never) to 4 (very often), full scale from 0-40, with higher score indicating higher perceived stress or the more often the person perceives stress.
Time Frame: Baseline and at 2-,4-, and 6-weeks
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline: number analyzed (Participants) | 13 | 12
  Baseline | 2.28 (0.34) | 2.36 (0.33)
  2 weeks: number analyzed (Participants) | 11 | 11
  2 weeks | 2.19 (0.35) | 2.17 (0.36)
  4 weeks: number analyzed (Participants) | 10 | 10
  4 weeks | 2.22 (0.35) | 2.28 (0.25)
  6 weeks: number analyzed (Participants) | 10 | 9
  6 weeks | 2.26 (0.41) | 2.18 (0.24)

6. Secondary Outcome: Change in Difficulty in Emotion Regulation Scale Scores (DERS)
Description: Difficulties in emotion regulation scale (DERS) The DERS is a 36-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 (" almost never [0-10%] ") to 5 (" almost always [91-100%] "). Total scale from 6-216. Higher scores indicate more difficulty in emotion regulation.
Time Frame: Baseline and at 2-,4-, and 6-weeks
Population: Results available for participants who completed instrument
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline: number analyzed (Participants) | 13 | 12
  Baseline | 119.15 (13.85) | 126.58 (19.66)
  2 weeks: number analyzed (Participants) | 11 | 11
  2 weeks | 109.09 (17.6) | 117.99 (17.80)
  4 weeks: number analyzed (Participants) | 10 | 10
  4 weeks | 110.2 (22.64) | 112.70 (30.67)
  6 weeks: number analyzed (Participants) | 10 | 9
  6 weeks | 104.07 (26.48) | 107.55 (29.06)

7. Secondary Outcome: Change in Beck Depression Scale Score (BDI)
Description: The Beck Depression Inventory (BDI) is used to evaluate depression symptoms. This questionnaire is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Scoring is from 0 (minimal) to 3 (severe), with total score from 0-63. Higher total scores indicate more severe depressive symptoms.
Time Frame: Baseline and at 2-,4-, and 6-weeks
Population: Data for participants who completed instrument
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline: number analyzed (Participants) | 13 | 12
  Baseline | 24.62 (9.45) | 20.08 (7.66)
  2 weeks: number analyzed (Participants) | 11 | 11
  2 weeks | 22.09 (10.55) | 15.36 (9.52)
  4 weeks: number analyzed (Participants) | 10 | 10
  4 weeks | 22.3 (14.02) | 16.3 (11.91)
  6 weeks: number analyzed (Participants) | 10 | 9
  6 weeks | 18.7 (13.26) | 16.67 (12.22)

8. Secondary Outcome: Change in State-Trait Anxiety Scale Score (STAXI)
Description: A 40 self-report items questionnaire, each item scored on 4-point likert-type response scale from 1 (not at all) to 4 (almost always), full range from 40 to 160, with higher score suggesting higher levels of anxiety.4
Time Frame: Baseline and at 2-,4-, and 6-weeks
Population: Data for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline: number analyzed (Participants) | 13 | 12
  Baseline | 84.54 (7.89) | 90.5 (8.72)
  2 weeks: number analyzed (Participants) | 11 | 11
  2 weeks | 86.91 (7.79) | 87.36 (8.08)
  4 weeks: number analyzed (Participants) | 10 | 10
  4 weeks | 90.9 (7.45) | 91.5 (9.41)
  6 weeks: number analyzed (Participants) | 10 | 9
  6 weeks | 90.7 (6.18) | 91.89 (8.87)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Cognitive Reappraisal-by-Distancing (CRD) | Control Downregulate Condition (CD)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT04967222/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT04967222/ICF_001.pdf